CLINICAL TRIAL: NCT04931147
Title: A Randomised, Double-blind, Placebo-controlled, SAD/MAD First-in-human, Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of RXC007 Including Evaluation of Drug-Drug Interaction and Food Effect in Male Participants
Brief Title: A 3-part Study to Evaluate Safety, Tolerability, Food Effect and Drug-drug Interactions of RXC007 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Redx Pharma Ltd (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RXC007/0001
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fibrosis; Inflammation; Idiopathic Pulmonary Fibrosis; Non-alcoholic Steatohepatitis; Liver Diseases; Kidney Diseases
MeSH Terms: conditions — Fibrosis; Inflammation; Idiopathic Pulmonary Fibrosis; Non-alcoholic Fatty Liver Disease; Liver Diseases; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This study is a first-in-human, single ascending (SAD) and multiple ascending dose (MAD) study, including the evaluation of drug-drug interactions. Each cohort will adopt a dose leader design with 2 participants being dosed on the first dosing day of each cohort. Of these 2, 1 will be on active drug and 1 on placebo. The remainder of the cohort will be dosed at least 24 h later pending an acceptable safety profile in the dose-leader group and will contain at least 1 additional placebo participant.
  In both Part A (SAD) and Part B (MAD), sequential cohorts will be exposed to increasing doses of RXC007. Prior to dose escalation between cohorts, safety and PK data from the previous cohort will be reviewed by the Dose Escalation Review Committee (DERC) to determine whether it is appropriate to proceed to the next cohort/dose level.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A & Part B of the study will assume a double blind design whereby both study participants and investigators will be blinded to active IMP versus placebo assignment. Within each cohort, 4 participants will be randomised to active versus 2 placebo participants.
  Part C of the study will assume an open-label design whereby all participants will receive active RXC007.
  A designated individual will generate the randomisation code under the guidance of a statistician. All other site and Sponsor personnel involved in the study will be blinded with regards to the IMP being administered. The Pharmacist (or designee) responsible for the preparation of participant doses and emergency code break envelopes will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Part A SAD - Cohort 1 (Experimental): This is the first treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive 2 mg of RXC007 on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Cohort 2 (Experimental): This is the second treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Cohort 1 Dose Escalation Data Review) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Cohort 3 (Experimental): This is the third treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Cohort 4 (Experimental): This is the fourth treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Cohort 5 (Experimental): This is the fifth treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Cohort 6 (Experimental): This is the sixth treatment arm in Part A (Single Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Optional Cohort 7 (Experimental): This is an optional seventh treatment arm in Part A (Single Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Optional Cohort 8 (Experimental): This is an optional eighth treatment arm in Part A (Single Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Cohort 1 (Experimental): This is the first treatment arm in Part B (Multiple Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of SAD cohort data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Cohort 2 (Experimental): This is the second treatment arm in Part B (Multiple Ascending Dose) of the study. 4 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of SAD and previous MAD cohort data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Optional Cohort 3 (Experimental): This is an optional third treatment arm in Part B (Multiple Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Optional Cohort 4 (Experimental): This is an optional fourth treatment arm in Part B (Multiple Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Optional Cohort 9 (Experimental): This is an optional ninth treatment arm in Part A (Single Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part A SAD - Optional Cohort 10 (Experimental): This is an optional tenth treatment arm in Part A (Single Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) on one occasion on Day 1. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Optional Cohort 5 (Experimental): This is an optional fifth treatment arm in Part B (Multiple Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part B MAD - Optional Cohort 6 (Experimental): This is an optional sixth treatment arm in Part B (Multiple Ascending Dose) of the study. If deemed as necessary following Dose Escalation Data Review of previous cohorts data, up to 8 participants may be enrolled into this optional cohort. If enrolled, up to 6 participants will be randomised to receive a selected dose of RXC007 (following Dose Escalation Data Review of previous cohorts data) once daily for 14 days. The remaining 2 participants will receive matching placebo.
  Interventions: Drug: RXC007; Drug: RXC007 Matching Placebo
- Part C DDI - Cohort 1 Rosuvastatin (Experimental): This is the first treatment arm in Part C (Drug-Drug Interaction) of the study. All participants within the cohort (12 participants) will to receive a selected dose of RXC007 (following Dose Escalation Data Review from Part A and Part B) and 10 mg rosuvastatin as follows: single dose of rosuvastatin (10 milligrams) on Day 1 followed by three single doses of RXC007 on Day 6, Day 7 & Day 8 before taking a single dose of both RXC007 and rosuvastatin together on Day 9.
  Interventions: Drug: RXC007
- Part C DDI - Cohort 2 Metformin (Experimental): This is the second treatment arm in Part C (Drug-Drug Interaction) of the study. All participants within the cohort (12 participants) will to receive a selected dose of RXC007 (following Dose Escalation Data Review from Part A and Part B) and 500 mg metformin as follows: single dose of metformin (500 milligrams) on Day 1 followed by three single doses of RXC007 on Day 4, Day 5 & Day 6 before taking a single dose of both RXC007 and metformin together on Day 7.
  Interventions: Drug: RXC007

INTERVENTIONS:
Drug: RXC007 — RXC007 will be administered in the form of oral capsules at selected doses starting at 2 mg to 4 of the 6 participants within each cohort in Part A and Part B. For Part A, dosing frequency is one single dose on one occasion and for Part B, dosing frequency is single doses once daily for 14 days. If required, following dose escalation data review, dosing frequency and duration may be modified in Part B.
  All participants in Part C (24) will receive active RXC007 in the form of oral capsules as single doses.
Drug: RXC007 Matching Placebo — The matching placebo for RXC007 will be administered in the form of oral capsules matched to the number of active RXC007 capsules at each dose level to 2 of the 6 participants within each cohort in Part A and Part B. For Part A, dosing frequency is one placebo dose on one occasion and for Part B, dosing frequency is single placebo doses once daily for 14 days. If required, following dose escalation data review, dosing frequency and duration may be modified in Part B.
  There is no placebo intervention for Part C of the study.
  Arms: Part A SAD - Cohort 1; Part A SAD - Cohort 2; Part A SAD - Cohort 3; Part A SAD - Cohort 4; Part A SAD - Cohort 5; Part A SAD - Cohort 6; Part A SAD - Optional Cohort 10; Part A SAD - Optional Cohort 7; Part A SAD - Optional Cohort 8; Part A SAD - Optional Cohort 9; Part B MAD - Cohort 1; Part B MAD - Cohort 2; Part B MAD - Optional Cohort 3; Part B MAD - Optional Cohort 4; Part B MAD - Optional Cohort 5; Part B MAD - Optional Cohort 6

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of RXC007.

DETAILED DESCRIPTION:
The study will be split into 3 parts: Part A, Part B & Part C.

The overall study will enrol up to 136 healthy males; maximum of 68 in Part A, maximum of 44 in Part B and maximum of 24 in Part C.

The purpose of Part A is to evaluate the safety, tolerability and concentration of RXC007 in the blood when it is given as a single dose on one occasion at different dose strengths. In addition, one group in Part A will investigate the effect of food on the safety, tolerability and concentration of RXC007 in the blood by taking a single dose of RXC007 following an overnight fast and then following a high fat breakfast. Part A will consist of 6 planned groups of 6 participants: each group investigating a different dose strength starting at the lowest dose and gradually increasing in each group. If required and determined as necessary following dose escalation data review, Part A may enrol up to a maximum of 4 additional cohorts with a maximum of 8 participants within each cohort.

Part A of the study will consist of a screening visit (between 28 and 2 days prior to first dose), a treatment period (consisting of a maximum of 5 days with 4 overnight stays) and a post-study follow-up visit on Day 15. For the food effect cohort, an additional treatment period (consisting of a maximum of 5 days with 4 overnight stays) will be undertaken following an approximately 4-week washout period with a second follow-up visit to be conducted on Day 15 following the second treatment period.

The purpose of Part B is to evaluate the safety, tolerability and concentration of RXC007 in the blood when it is given as a single dose once a day for a period of 14 days at different dose strengths. Part B will consist of up to 2 planned groups of 6 participants; each group investigating a different dose strength based on the data generated during Part A of the study. If required and determined as necessary following dose escalation data review, Part B may enrol up to a maximum of 4 additional cohorts with a maximum of 8 participants within each cohort.

Part B of the study will consist of a screening visit (between 28 and 2 days prior to first dose), a treatment period (consisting of a maximum of 18 days with 17 overnight stays) and a post-study follow-up visit on Day 28.

Within each cohort in Part A and Part B, 4 participants will receive RXC007 with the remaining 2 participants receiving a matching placebo. Each cohort will follow a dose leader schedule, whereby 2 participants (1 active, 1 placebo) will be dosed a minimum of 24 hours prior to the remaining 4 participants in the cohort. Between each cohort, safety and PK data up to the 72-hour post-last dose time point for Part A and up to Day 17 in Part B will be evaluated by a Dose Escalation Review Committee (DERC) to determine whether it is appropriate to dose escalate into the next cohort. If required, i.e., the safety or pharmacokinetics (PK) data indicates, dose modifications may be made in order to select an intermediate/lower dose. In addition, modifications may be made following both treatment periods for the food effect cohort in Part A to dose all remaining cohorts in Part A and Part B in a fed state (with a standardised breakfast) and in Part B, the dose regime may be modified in terms of frequency to increase dosing from once per day to multiple times per day. In addition, decisions may be made that the proposed length of the in-house treatment period in both Part A & Part B should be reduced by one day (from Day 4 to Day 3 in Part A and from Day 17 to Day 16 in Part B).

The purpose of Part C is to evaluate the safety, tolerability and effect of RXC007 on the concentration of rosuvastatin and metformin in the blood to determine as to whether RXC007 affects the activity of the processes by which certain types of drugs are broken down (metabolised) in the body and therefore, whether RXC007 has the potential to interact with other drugs, affecting their desired effect in the body i.e., evaluating the drug-drug interaction potential of RXC007.

Part C will consist of 2 groups of 12 participants; Group 1 evaluating the drug-drug interactions of RXC007 and rosuvastatin (at a dose strength of 10 mg in an oral tablet formulation) and Group 2 evaluating the drug-drug interactions of RXC007 and metformin (at a dose strength of 500 mg in an oral tablet formulation). The dose strength of RXC007 to be evaluated will be selected based on review of the data generated in Part B of the study.

Part C of the study will consist of a screening visit (between 28 and 2 days prior to first dose), a treatment period (consisting of either a maximum of 14 days with 13 overnight stays for Group 1 or a maximum of 11 days with 10 overnight stays for Group 2) and a post-study follow-up visit approximately 14 days following the last dose of RXC007 with rosuvastatin or metformin (either Day 23 or Day 21 respectively for Group 1 and Group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male participants, between 18 and 55 years of age, inclusive.
2. Male participant (and female partner of childbearing potential) willing to use a highly effective method of contraception or 2 effective methods of contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the participant) from first dose until 3 months after last dose of IMP/NIMP.
3. Participant with a body mass index (BMI) of 18.0-32.0 kg/m2.
4. Participant with a body weight of 60 kg or greater.
5. No clinically significant history of previous allergy / sensitivity to RXC007, rosuvastatin or metformin, or any of the excipients contained within the IMP/NIMP.
6. No clinically significant abnormal test results for serum biochemistry, haematology and/or urine analyses within 28 days before the first dose administration of the IMP/NIMP.
7. Haemoglobin and haematocrit above the lower limit of the normal range for the reference laboratory.
8. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 1.5 times the upper limit of the normal (ULN) range for the reference laboratory.
9. Participant with a negative urinary drugs of abuse (DOA) screen (including alcohol) test results, determined within 28 days before the first dose administration of the IMP/NIMP (N.B.: A positive test result may be repeated at the Investigator's discretion).
10. Participant with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) test results at Screening.
11. No clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before first dose of IMP/NIMP including a PR interval > 220ms, QRS width > 120ms and QTcF interval > 450 ms.
12. No clinically significant abnormalities in vital signs (e.g., blood pressure (systolic blood pressure > 140 mmHg) / heart rate, respiration rate, oral temperature) determined within 28 days before first dose of IMP/NIMP.
13. Participant must be available to complete the study (including all follow-up visits).
14. Participant must satisfy an Investigator about his fitness to participate in the study.
15. Participant must provide written informed consent to participate in the study.
16. Participants with a negative COVID-19 reverse transcription polymerase chain reaction (RT-PCR) test on admission (if required).

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence IMP/NIMP absorption.
2. A clinically significant history of infection in the last 3 months.
3. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements, antacids (Part C Cohort 1 only), any product known to be a substrate mainly metabolised by CYP enzymes within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMP/NIMP.
4. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
5. Participants who are unable to demonstrate the ability to swallow multiple "dummy" capsules (i.e., an empty gelatin capsules) of the size proposed for administration in a particular cohort/dose level (up to and including size 00).
6. Participant with a glomerular filtration rate less than 80 mL/min/1.73m2 (calculated by Cockcroft-Gault equation.
7. A clinically significant history of drug or alcohol abuse (defined as the consumption of more than 14 units of alcohol a week) within the past two years.
8. Inability to communicate well with the Investigators (i.e., language problem, poor mental development or impaired cerebral function).
9. Participation in a NCE clinical study within the previous 3 months or five half-lives, whichever is longer, or a marketed drug clinical study within the 30 days or five half-lives, whichever is longer, before the first dose of IMP/NIMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
10. Donation of 450 mL or more blood within the 3 months before the first dose of IMP/NIMP.
11. Vegans, vegetarians or other dietary restrictions (e.g., restrictions for medical, religious or cultural reasons, etc.), which would prevent participants from consuming a high-fat breakfast or standardised meal.
12. Users of nicotine products i.e., current smokers or ex-smokers who have smoked within the 6 months prior to screening or users of cigarette replacements (i.e., e-cigarettes, nicotine patches or gums).
13. Participants who have received a COVID-19 vaccine injection within 28 days prior to the first dose of IMP/NIMP.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As this is a first-in-human (FiH) study, as per the EMA guidance for risk mitigation in FiH studies, the most relevant population is healthy male volunteers.
Enrollment: 90 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | Collection of TEAEs occurs through ad hoc reporting from the participants from the point of first dose administration (Day 1 in each part) through to study completion (up to 6 weeks for Part A & up to 8 weeks for Part B & C).
  This primary endpoint relates to the number of participants who report a treatment emergent adverse event (TEAEs) across all study parts.
Number of participants who report a change from normal range values for laboratory safety parameters (serum biochemistry, serum haematology or urinalysis) from first dose on Day 1 to post-study follow up visit. | Part A: From Day 1 to post-study follow up visit (up to 6 weeks) & Part B/C: From Day 1 to post-study follow up visit (up to 8 weeks)
  This primary endpoint will report the number of participants within each cohort of Part A, Part B & Part C of the study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the serum biochemistry, serum haematology or urinalysis parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the post-study visit.
Number of participants who report a change from normal range values for vital signs parameters (blood pressure, pulse rate, respiration rate, oral body temperature) from first dose on Day 1 to post-study follow up visit. | Part A: From Day 1 to post-study follow up visit (up to 6 weeks) & Part B/C: From Day 1 to post-study follow up visit (up to 8 weeks)
  This primary endpoint will report the number of participants within each cohort of Part A, Part B & Part C of the study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the vital signs parameters (systolic/diastolic blood pressure, pulse rate, respiration rate, oral body temperature) as defined in the study protocol following first dose administration on Day 1 up to completion of the post-study visit.
Number of participants who report a change from normal range values for any of the associated 12-Lead ECG parameters (heart rate, PR interval, QRS width, QT interval and QTcF interval) from first dose on Day 1 to post-study follow up visit. | Part A: From Day 1 to post-study follow up visit (up to 6 weeks) & Part B/C: From Day 1 to post-study follow up visit (up to 8 weeks)
  This primary endpoint will report the number of participants within each cohort of Part A, Part B & Part C of the study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the 12-Lead ECG parameters (heart rate, PR interval, QRS width, QT interval and QTcF interval) as defined in the study protocol following first dose administration on Day 1 up to completion of the post-study visit.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters - Part A - Maximum observed concentration (Cmax) | Plasma samples for Cmax evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the maximum observed concentration (Cmax) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Time to maximum observed concentration (Tmax) | Plasma samples for Tmax evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the time to maximum observed concentration (Tmax) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Elimination rate constant (λz) | Plasma samples for λz evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the elimination rate constant (λz) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Terminal elimination half-life (t1/2) | Plasma samples for t1/2 evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the terminal elimination half-life (t1/2) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) | Plasma samples for AUC0-t evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) | Plasma samples for AUC0-inf evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Residual Area (AUC%extrapolated) | Plasma samples for AUC%extrapolated evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the residual area (AUC%extrapolated) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Total apparent clearance following extravascular administration (CL/F) | Plasma samples for CL/F evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the total apparent clearance following extravascular administration (CL/F) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part A - Apparent volume of distribution following extravascular administration (Vz/F) | Plasma samples for Vz/F evaluation of RXC007 in Part A: Day 1 pre-dose, 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, 48 hr, 72 hr post-dose & post-study follow up (up to 6 weeks for Part A).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the apparent volume of distribution following extravascular administration (Vz/F) of RXC007 in plasma for Part A cohorts.
Pharmacokinetic Parameters - Part B - Maximum observed concentration (Cmax) | Plasma samples for Cmax evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the maximum observed concentration (Cmax) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Time to maximum observed concentration (Tmax) | Plasma samples for Tmax evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the time to maximum observed concentration (Tmax) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Elimination rate constant (λz) | Plasma samples for λz evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the elimination rate constant (λz) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Terminal elimination half-life (t1/2) | Plasma samples for t1/2 evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the terminal elimination half-life (t1/2) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Area under the concentration-time curve (AUC) from 0 to τ, where τ is the dosing interval (0 - 24 h) (AUC0-τ) | Plasma samples for AUC0-τ evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) from 0 to τ, where τ is the dosing interval (0 - 24 h) (AUC0-τ) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) | Plasma samples for AUC0-t evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) | Plasma samples for AUC0-inf evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Residual area (AUC%extrapolated) | Plasma samples for AUC%extrapolated evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the residual area (AUC%extrapolated) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Accumulation ratio calculated from Cmax (ARCmax) | Plasma samples for ARCmax evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the accumulation ratio calculated from Cmax (ARCmax) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Accumulation ratio calculated from AUC (ARAUC) | Plasma samples for ARAUC evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the accumulation ratio calculated from AUC (ARAUC) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Total apparent clearance following extravascular administration (CL/F) | Plasma samples for CL/F evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the total apparent clearance following extravascular administration (CL/F) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part B - Apparent volume of distribution following extravascular administration (Vz/F) | Plasma samples for Vz/F evaluation of RXC007 in Part B: Day 1 & 14: 15 mins, 30 mins, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr post-dose, Day 7, Day 16: 48 hr post-Day 14 dose & Day 17: 72 hr post-Day 14 dose (up to 8 weeks for Part B).
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the apparent volume of distribution following extravascular administration (Vz/F) of RXC007 in plasma for Part B cohorts.
Pharmacokinetic Parameters - Part C - Maximum observed concentration (Cmax) | Plasma samples for Cmax evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the maximum observed concentration (Cmax) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Time to maximum observed concentration (Tmax) | Plasma samples for Tmax evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the time to maximum observed concentration (Tmax) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Elimination rate constant (λz) | Plasma samples for λz evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the time to elimination rate constant (λz) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Terminal elimination half-life (t1/2) | Plasma samples for t1/2 evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the time to terminal elimination half-life (t1/2) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) | Plasma samples for AUC0-t evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration (AUC0-t) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) | Plasma samples for AUC0-inf evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Residual area (AUC%extrapolated) | Plasma samples for AUC%extrapolated evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the residual area (AUC%extrapolated) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Total apparent clearance following extravascular administration (CL/F) | Plasma samples for CL/F evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the total apparent clearance following extravascular administration (CL/F) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.
Pharmacokinetic Parameters - Part C - Apparent volume of distribution following extravascular administration (Vz/F) | Plasma samples for Vz/F evaluation of in Part C: Maximum of 34 samples in Cohort 1 from Day 1 pre-dose to Day 13 and maximum of 33 samples in Cohort 2 from Day 1 pre-dose to Day 10
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007, Rosuvastatin and Metformin. This endpoint will report the summary of derived pharmacokinetic parameters for the apparent volume of distribution following extravascular administration (Vz/F) of RXC007, rosuvastatin and metformin in plasma for Part C cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, Principal Investigator — Simbec-Orion Clinical Pharmacology
Locations (1):
- Simbec-Orion Clinical Pharmacology, Merthyr Tydfil, Mid Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At this stage, it is not planned that any IPD information will be shared with other researchers outside of the Sponsor and Clinical Research Organisation undertaking the conduct of this study.